CLINICAL TRIAL: NCT02624947
Title: A Phase 3, Randomized, Observer-Blind, Placebo-Controlled, Group-Sequential Study to Determine the Immunogenicity and Safety of a Respiratory Syncytial Virus (RSV) F Nanoparticle Vaccine With Aluminum in Healthy Third-trimester Pregnant Women; and Safety and Efficacy of Maternally Transferred Antibodies in Preventing RSV Disease in Their Infants
Brief Title: A Study to Determine the Safety and Efficacy of the RSV F Vaccine to Protect Infants Via Maternal Immunization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RSV-M-301
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group A (Placebo Comparator): Formulation buffer (0.5mL injection)
  Interventions: Biological: Formulation buffer
- Treatment Group (Active Comparator): RSV F vaccine with adjuvant (0.5mL injection)
  Interventions: Biological: RSV F vaccine with adjuvant

INTERVENTIONS:
Biological: RSV F vaccine with adjuvant
  Arms: Treatment Group
Biological: Formulation buffer
  Arms: Treatment Group A

SUMMARY:
The purpose of this study is to determine the efficacy of maternal immunization during the third trimester of pregnancy with the RSV F vaccine against medically-significant RSV lower respiratory tract infection (LRTI), as defined by hypoxemia or tachypnea at rest, through the first 90, 120, 150, and 180 days of life in infants.

DETAILED DESCRIPTION:
This is a randomized, observer-blind, placebo-controlled trial enrolling third-trimester pregnant women in the Northern and Southern hemispheres, for up to four consecutive RSV seasons in each hemisphere. The trial could enroll up to 8618 third-trimester pregnant subjects, of which 4,636 were actually enrolled. Women in the third trimester of a singleton uncomplicated low-risk pregnancy and 18 to 40 years of age (inclusive) were enrolled and randomized in a 1:1 ratio into one of two treatment groups, active or placebo, over approximately three months prior to peak RSV season in their locale. After the first global season of enrollment, the randomization scheme was changed to a 2:1 (active/placebo) ratio to enable a more efficient accrual of the safety database.

All maternal subjects were to receive a single intramuscular (IM) injection on Day 0 with the assigned test article, the RSV F vaccine, or placebo. Study participation for maternal subjects spanned approximately nine (9) months from the first dose, ending six (6) months post-delivery. Study follow-up for live-born infant subjects spanned approximately one (1) year post-delivery.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤40 years-of-age
2. Singleton pregnancy of 28 to 36 0/7 weeks gestation on the day of planned vaccination

   * Documentation of gestational age will be based on one of the following composite criteria. (Note: The Investigator was to use the earliest ultrasound data available to establish the study-specific gestational age dating):

     1. Gestational Age Dating Based on First Trimester Data (data obtained ≤13 6/7 weeks): The date of the first day of the reported last menstrual period (LMP) may be used to establish the gestational age if corroborated by a first trimester ultrasound. If the gestational age estimation derived using the LMP and the first trimester ultrasound are discrepant >7 days, the ultrasound will be used to establish gestational age. If LMP is uncertain or unknown, the ultrasound-established gestational age estimation will be used to establish the gestational age of the pregnancy.
     2. Gestational Age Dating Based on Early Second Trimester Data (data obtained 14 0/7 to 21 6/7 weeks): The day of the first reported LMP may be used to establish the gestational age if corroborated by an early second trimester ultrasound (that estimates the gestational age between 14 0/7 and 21 6/7 weeks). If the gestational age estimation derived using the LMP and the early second trimester ultrasound are discrepant >10 days, the ultrasound will be used to establish the gestational age. If LMP is uncertain or unknown, the ultrasound-established gestational age estimation will be used to establish the gestational age of the pregnancy.
     3. Gestation Age Dating Based on Later Second Trimester Data (data obtained 22 0/7 and 27 6/7 weeks by LMP): The date of the first day of the reported LMP may be used to establish the gestation age if corroborated by a later second trimester ultrasound (that estimates the gestational age between 22 0/7 and 27 6/7 weeks). If the gestational age estimation derived using the LMP and the later second trimester ultrasound are discrepant >14 days, the ultrasound will be used to establish the gestational age. If LMP is uncertain or unknown, the ultrasound-established gestational age estimation will be used to establish the gestational age of the pregnancy.
     4. Gestational Age Dating When the LMP is Uncertain or Unknown AND No Prior First or Second Trimester Ultrasound Has Been Performed: An ultrasound performed at screening within the second trimester (≤27 6/7 weeks) will be used to establish the gestational age of the pregnancy.
3. Documentation of a second or third (between 18 0/7 weeks and prior to randomization) trimester ultrasound with no major fetal anomalies identified.
4. Good general maternal health as demonstrated by:

   * Medical history (including history of adverse reactions to prior vaccines and allergies).
   * Physical examination including at least vital signs (blood pressure, pulse, respirations, and oral temperature); weight; height; examination of the HEENT, cardiovascular, pulmonary, gastrointestinal (abdominal), musculoskeletal, lymphatic, and dermatologic organ systems; and documentation of fetal heart tones. Note that abnormal vital signs may be repeated at the investigator's discretion since these measures may be labile. Vital signs should be assessed in the context of normal values for the third trimester of pregnancy (see the Study Operations Manual).
   * Clinical laboratory parameters that include:

     * For the first year of study conduct in any country, normal/clinically insignificant blood urea nitrogen (BUN), creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase (ALP), hemoglobin, white blood count, and platelet count. Note that normal ranges for clinical laboratory parameters will be based on reference ranges appropriate for the subject population under study (i.e., third trimester of pregnancy) and as defined in the toxicity grading scale (TGS) (see the Study Operations Manual).
     * For all subjects, serologic exclusion of infection with hepatitis B (HBV) and C (HCV) viruses, syphilis, and HIV as documented by testing (performed at the central or local laboratory) at screening or by medical records during the current pregnancy.
5. Able to understand, and both willing and physically able to comply with study procedures. This includes anticipation of reasonable geographic proximity to the study clinic and adequate transportation to comply with scheduled and unscheduled study follow-up visits.
6. Able and willing to provide written informed consent for themselves and infant.

Exclusion Criteria:

1. Symptomatic cardiac or pulmonary disease requiring chronic drug therapy, including hypertension and asthma. Asthma will be exclusionary if the subject is receiving chronic systemic glucocorticoids at any dose or inhaled glucocorticoids at any dose >500µg per day of beclomethasone or fluticasone, or >800μg per day of budesonide.
2. Pregnancy complications (in the current pregnancy) such as preterm labor, hypertension (blood pressure [BP] >140/90 in the presence of proteinuria or BP >150/100 with or without proteinuria) or currently on an antihypertensive therapy or pre-eclampsia; or evidence of intrauterine growth restriction.
3. Grade 2 or higher clinical laboratory or vital sign abnormality. Exclusion of subjects with grade 1 abnormalities will be based on the subject's prior medical history and the investigator's clinical judgment that the abnormality is indicative of a meaningful physiologic event.
4. Receipt of any licensed vaccine (e.g., Tdap, inactivated influenza vaccine) within 14 days of study vaccination.
5. Received any RSV vaccine at any time.
6. Body mass index (BMI) of ≥40, at the time of the screening visit.
7. Hemoglobinopathy (even if asymptomatic) or blood dyscrasias.
8. Hepatic or renal dysfunction.
9. Established diagnosis of seizure disorder, regardless of therapy.
10. Known, active auto-immune disease or immunodeficiency syndrome.
11. Endocrine disorders, including (but not limited to) untreated hyperthyroidism, untreated hypothyroidism (unless due to auto-immune disease), and glucose intolerance (e.g., diabetes mellitus type 1 or 2) antedating pregnancy, or occurring during pregnancy and requiring interventions other than diet for control.
12. History of major gynecologic or major abdominal surgery, including bariatric surgery (previous Caesarean section is not an exclusion).
13. Known HIV, syphilis, HBV, or HCV infection, as assessed by serologic tests conducted during the current pregnancy or as a procedure during the screening period of the study.
14. Primary genital Herpes simplex virus (HSV) infection during the current pregnancy.
15. Current alcohol or drug abuse based on the Investigator's knowledge of present or recent (within the last 2 years) use/abuse of alcohol or illegal or non-prescription drugs.
16. Documentation that the current pregnancy results from in vitro fertilization (IVF).
17. Documentation that the current pregnancy results from rape or incest.
18. Documentation that the infant will be a ward of the state or be released for adoption.
19. History/presence of deep venous thrombosis or thromboembolism, or the use of anticoagulants during pregnancy (the use of low-dose aspirin as prophylaxis [e.g., for the prevention of morbidity and mortality from preeclampsia] is acceptable is dosages consistent with local standards of care).
20. Red blood cell allo-immunization.
21. Prior stillbirth or neonatal death, or multiple (≥3) spontaneous abortions.
22. Prior preterm delivery ≤34 weeks gestation or having ongoing intervention (medical/surgical) in current pregnancy to prevent preterm birth.
23. Greater than five (5) prior deliveries.
24. Previous infant with a known genetic disorder or major congenital anomaly.
25. Receipt of investigational drugs or immune globulins (with the exception of prophylactic anti-Rho D immune globulin) within six (6) months prior to the administration of the study vaccine.
26. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted except for the limit established in exclusion criterion #1.
27. Neuro-psychiatric illness deemed likely to interfere with protocol compliance, safety reporting, or receipt of pre-natal care; or requiring treatment with psychotropic drugs (excluding treatment for depression and anxiety).
28. Any other physical, psychiatric or social condition which may, in the investigator's opinion, increase the risks of study participation to the maternal subject or the fetus/infant; or may lead to the collection of incomplete or inaccurate safety data.
29. Acute disease within 72 hours of the day of the planned vaccination (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C).
30. History of a serious adverse reactions (e.g., anaphylaxis) to any prior vaccine.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4636 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12-28 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax Inc
Locations (88):
- United States (49):
  - Research Site US115, Birmingham, Alabama
  - Research Site US035, Cullman, Alabama
  - Research Site US130, Fort Defiance, Arizona
  - Research Site US123, Phoenix, Arizona
  - Research Site US103, Tucson, Arizona
  - Research Site US129, Whiteriver, Arizona
  - Research Site US092, Colton, California
  - Research Site US114, Huntington Park, California
  - Research Site US127, Los Angeles, California
  - Research Site US091, Madera, California
  - Research Site US093, Riverside, California
  - Research Site US134, Aurora, Colorado
  - Research Site US036, Denver, Colorado
  - Research Site US040, Washington D.C., District of Columbia
  - Research Site US037, Blackfoot, Idaho
  - Research Site US119, Idaho Falls, Idaho
  - Research Site US032, Nampa, Idaho
  - Research Site US095, Chicago, Illinois
  - Research Site US090, West Des Moines, Iowa
  - Research Site US038, Augusta, Kansas
  - Research Site US031, Hutchinson, Kansas
  - Research Site US096, Louisville, Kentucky
  - Research Site US126, Alexandria, Louisiana
  - Research Site US039, Metairie, Louisiana
  - Research Site US101, Detroit, Michigan
  - Research Site US098, Biloxi, Mississippi
  - Research Site US102, Lincoln, Nebraska
  - Research Site US025, Norfolk, Nebraska
  - Research Site US088, Neptune City, New Jersey
  - Research Site US131, Gallup, New Mexico
  - Research Site US087, Johnson City, New York
  - Research Site US086, Syracuse, New York
  - Research Site US020, Durham, North Carolina
  - Research Site US097, Fort Bragg, North Carolina
  - Research Site US089, Englewood, Ohio
  - Research Site US021, Pittsburgh, Pennsylvania
  - Research Site US116, Beaumont, Texas
  - Research Site US083, Fort Worth, Texas
  - Research Site US043, Galveston, Texas
  - Research Site US019, Houston, Texas
  - Research Site US128, Houston, Texas
  - Research Site US125, Lampasas, Texas
  - Research Site US094, Longview, Texas
  - Research Site US042, San Antonio, Texas
  - Research Site US121, Salt Lake City, Utah
  - Research Site US008, Salt Lake City, Utah
  - Research Site US099, Salt Lake City, Utah
  - Research Site US100, Richmond, Virginia
  - Research Site US041, Seattle, Washington
- Argentina (5):
  - Research Site AR002, Buenos Aires
  - Research Site AR006, Córdoba
  - Research Site AR011, Mendoza
  - Research Site AR008, Salta
  - Research Site AR003, San Miguel de Tucumán
- Australia (5):
  - Research Site AU010, Brisbane, Queensland
  - Research Site AU007, Adelaide, South Australia
  - Research Site AU011, Clayton, Victoria
  - Research Site AU008, Melbourne, Victoria
  - Research Site AU009, Perth, Western Australia
- Research Site BD001, Sylhet, Sylhet Division, Bangladesh
- Chile (3):
  - Research Site CL002, Osorno, Los Lagos Region
  - Research Site CL001, Santiago, Region Metropolitana (RM)
  - Research Site CL003, Concepción, Región del Biobío
- Research Site MX001, Monterrey, Nuevo León, Mexico
- New Zealand (4):
  - Research Site NZ003, Grafton, Auckland
  - Research Site NZ001, Papatoetoe, Aukland
  - Research Site NZ002, Christchurch
  - Research Site NZ004, Wellington
- Philippines (2):
  - Research Site PH001, Alabang, Manila
  - Research Site PH002, Muntinlupa, National Capital Region
- South Africa (10):
  - Research Site ZA004, Parow, Cape Town
  - Research Site ZA003, Hillbrow, Johannesburg
  - Research Site ZA007, Thabazimbi, Limpopo Providence
  - Research Site ZA010, Bellville, Western Cape
  - Research Site ZA009, Paarl, Western Cape
  - Research Site ZA011, Worcester, Western Cape
  - Research Site ZA006, Benoni
  - Research Site ZA008, Bloemfontein
  - Research Site ZA002, Soshanguve
  - Research Site ZA001, Soweto
- Spain (4):
  - Research Site ES002, Barcelona
  - Research Site ES003, Madrid
  - Research Site ES004, Santiago de Compostela
  - Research Site ES001, Seville
- United Kingdom (4):
  - Research Site UK004, Bristol
  - Research Site UK001, London
  - Research Site UK002, Oxford
  - Research Site UK003, Southampton

REFERENCES:
- [Derived] Madhi SA, Polack FP, Piedra PA, Munoz FM, Trenholme AA, Simoes EAF, Swamy GK, Agrawal S, Ahmed K, August A, Baqui AH, Calvert A, Chen J, Cho I, Cotton MF, Cutland CL, Englund JA, Fix A, Gonik B, Hammitt L, Heath PT, de Jesus JN, Jones CE, Khalil A, Kimberlin DW, Libster R, Llapur CJ, Lucero M, Perez Marc G, Marshall HS, Masenya MS, Martinon-Torres F, Meece JK, Nolan TM, Osman A, Perrett KP, Plested JS, Richmond PC, Snape MD, Shakib JH, Shinde V, Stoney T, Thomas DN, Tita AT, Varner MW, Vatish M, Vrbicky K, Wen J, Zaman K, Zar HJ, Glenn GM, Fries LF; Prepare Study Group. Respiratory Syncytial Virus Vaccination during Pregnancy and Effects in Infants. N Engl J Med. 2020 Jul 30;383(5):426-439. doi: 10.1056/NEJMoa1908380. PMID 32726529
- See also: Novavax, Inc — http://novavax.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in a study at 86 sites in 11 different countries from 03 December 2015 to 12 July 2019.
Pre-assignment Details: Healthy women 18-40 years of age with low-risk singleton pregnancies enrolled and treated in the study with 120 µg Respiratory Syncytial Virus Recombinant F (RSVF) nanoparticle vaccine adsorbed to 0.4 mg of Aluminum (as phosphate salt) ) or formulated buffer (placebo control) as a single 0.5 mL IM (Intramuscular) injection into the deltoid muscle.
Groups:
- Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum): Maternal participants were administered with the adjuvanted RSV F vaccine 120 µg RSV F protein adsorbed to a 0.4 mg dose of aluminum (as the phosphate salt) as a single 0.5 mL IM injection into the deltoid muscle.
- Formulated Buffer (Placebo Control): Maternal participants were administered with the formulated buffer (placebo control) as a single 0.5 mL IM injection into the deltoid muscle.
Period: Maternal Participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Started | 3051 | 1585
Participants in Safety Population | 3045 | 1581
Completed | 2907 | 1510
Not Completed | 144 | 75
Not completed — Adverse Event | 5 | 0
Not completed — Investigator Decision | 5 | 3
Not completed — Lost to Follow-up | 54 | 24
Not completed — Non Compliance | 8 | 5
Not completed — Sponsor Request | 1 | 1
Not completed — Voluntary withdrawal unrelated to AE | 48 | 27
Not completed — Miscellaneous | 23 | 15
Period: Infant Participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Started | 3014 | 1565
Participants in Safety Population | 3008 | 1561
All Live Births | 3014 | 1565
Completed | 2783 | 1433
Not Completed | 231 | 132
Not completed — Adverse Event | 18 | 11
Not completed — Investigator Decision | 5 | 4
Not completed — Lost to Follow-up | 93 | 58
Not completed — Non Compliance | 17 | 7
Not completed — Sponsor Request | 0 | 1
Not completed — Voluntary Withdrawal unrelated to AE | 48 | 25
Not completed — Miscellaneous | 50 | 26

BASELINE CHARACTERISTICS:
Population: The maternal safety population (S-M) included all maternal participants who received any test article and were analyzed as randomized unless conclusive documentation existed to confirm the mis-dosing of a maternal subject and the identity of the treatment actually received.
  The infant safety population (S-I) included the infants of maternal subjects who received any test article.
Groups:
- Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum): Maternal participants were administered the adjuvant RSV F vaccine (120 µg RSV F protein adsorbed to a 0.4 mg dose of aluminum as the phosphate salt) as a single 0.5 mL IM injection into the deltoid muscle.
  Infants were monitored and data was collected based on the intervention given to the mothers.
- Formulated Buffer (Placebo Control): Maternal participants were administered the formulated buffer (placebo control) as a single 0.5 mL IM injection into the deltoid muscle. Infants were monitored and data was collected based on the intervention given to the mothers.
- Total: Total of all reporting groups
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control) | Total
Number analyzed (Participants) | 3045 | 1581 | 4626
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5.3) | 26 (5.2) | 26 (5.3)
Age, Customized [Mean (Standard Deviation); unit: weeks] — Population: Analysis population includes infant participants who were ≥ 37 weeks GA at birth, and born to maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery, and had not received prophylactic treatment with palivizumab between birth and Day 180 after delivery, and had at least 1 documented post-partum contact during which active and/or passive surveillance activities for RSV-suspect illness could occur.
  weeks
    Gestational Age at delivery (Infant Population): number analyzed (Participants) | 3008 | 1561 | 4569
    Gestational Age at delivery (Infant Population) | 39.3 (1.49) | 39.3 (1.58) | 39.3 (1.52)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3045 | 1581 | 4626
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Analysis population includes infant participants who were ≥ 37 weeks GA at birth, and born to maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery, and had not received prophylactic treatment with palivizumab between birth and Day 180 after delivery, and had at least 1 documented post-partum contact during which active and/or passive surveillance activities for RSV-suspect illness could occur.
  Participants
    Male: number analyzed (Participants) | 3008 | 1561 | 4569
    Male | 1556 | 799 | 2355
    Female: number analyzed (Participants) | 3008 | 1561 | 4569
    Female | 1449 | 757 | 2206
    No data: number analyzed (Participants) | 3008 | 1561 | 4569
    No data | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 409 | 212 | 621
  Not Hispanic or Latino | 2636 | 1369 | 4005
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 11 | 33
  Asian | 320 | 168 | 488
  Native Hawaiian or Other Pacific Islander | 49 | 27 | 76
  Black or African American | 1335 | 682 | 2017
  White | 903 | 489 | 1392
  More than one race | 416 | 204 | 620
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Analysis population includes infant participants who were ≥ 37 weeks GA at birth, and born to maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery, and had not received prophylactic treatment with palivizumab between birth and Day 180 after delivery, and had at least 1 documented post-partum contact during which active and/or passive surveillance activities for RSV-suspect illness could occur.
  Participants
    White or Caucasian: number analyzed (Participants) | 3008 | 1561 | 4569
    White or Caucasian | 900 | 477 | 1377
    Black or African American: number analyzed (Participants) | 3008 | 1561 | 4569
    Black or African American | 1387 | 696 | 2083
    Asian: number analyzed (Participants) | 3008 | 1561 | 4569
    Asian | 310 | 162 | 472
    American Indian or Alaska Native: number analyzed (Participants) | 3008 | 1561 | 4569
    American Indian or Alaska Native | 21 | 9 | 30
    Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 3008 | 1561 | 4569
    Native Hawaiian or other Pacific Islander | 55 | 28 | 83
    Other: number analyzed (Participants) | 3008 | 1561 | 4569
    Other | 333 | 187 | 520
    No data: number analyzed (Participants) | 3008 | 1561 | 4569
    No data | 2 | 2 | 4
    Hispanic or Latino: number analyzed (Participants) | 3008 | 1561 | 4569
    Hispanic or Latino | 403 | 213 | 616
    Not Hispanic or Latino: number analyzed (Participants) | 3008 | 1561 | 4569
    Not Hispanic or Latino | 2603 | 1346 | 3949
    Na data: number analyzed (Participants) | 3008 | 1561 | 4569
    Na data | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Infants: Percentages of Participants With Medically Significant RSV LRTI With Either Hypoxemia (SpO2 <95% at Sea Level or <92% at Altitudes >1800 Meters) or Tachypnea
Description: Percentages of infants with medically-significant RSV LRTI from delivery through 90, 120,150, and 180 days of life, as defined by:
  * The presence of RSV infection confirmed by detection of RSV genome by RT-PCR on respiratory secretions (obtained within the continuous illness episode which fulfills the other criteria listed below); AND
  * At least one manifestation of lower respiratory tract infection (LRTI) from among the following: cough, nasal flaring, lower chest wall indrawing, subcostal retractions, stridor, rales, rhonchi, wheezing, crackles/crepitations, or observed apnea; AND
  * Evidence of medical significance as defined by the presence of:
    * EITHER hypoxemia (peripheral oxygen saturation [SpO2] < 95% at sea level or < 92% at altitudes > 1800 meters) OR
    * Tachypnea (≥ 70 breaths per minute [bpm] in infants 0 to 59 days of age and ≥ 60 bpm in infants ≥ 60 days of age).
Time Frame: Delivery to 180 days after delivery
Population: Analysis population includes infant participants who were ≥ 37 weeks GA at birth, and born to maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery, and had not received prophylactic treatment with palivizumab between birth and Day 180 after delivery, and had at least 1 documented post-partum contact during which active and/or passive surveillance activities for RSV-suspect illness could occur.
Measure: Count of Participants; unit: Participants
Groups:
- Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum): Maternal participants were administered with the adjuvanted RSV F vaccine (120 µg RSV F protein adsorbed to a 0.4 mg dose of aluminum as the phosphate salt) as a single 0.5 mL IM injection into the deltoid muscle.
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 2765 | 1430
Participants
  Day 90 | 41 | 35
  Day 120 | 52 | 41
  Day 150 | 57 | 43
  Day 180 | 61 | 43

2. Secondary Outcome: Infants: Number of Participants With RSV LRTI With Severe Hypoxemia (Sp02 <92% at Sea Level or <87% at Altitudes >1800 Meters) or Documented Use of Oxygen by High Flow Nasal Cannula or Other Advanced Respiratory Support Through 90 Days of Life
Description: The number of infants with RSV LRTI with EITHER severe hypoxemia (SpO2 < 92% at sea level or < 87% at altitudes > 1800 meters) OR the documented use of oxygen by high flow nasal cannula OR CPAP OR BiPAP OR Bubble CPAP OR bag-mask ventilation OR intubation with subsequent mechanical (or manual) ventilation OR ECMO from delivery through 90, 120, 150, and 180 days of life.
Time Frame: Delivery to 180 days after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 2765 | 1430
Participants
  Day 90 | 14 | 14
  Day 120 | 16 | 16
  Day 150 | 17 | 17
  Day 180 | 19 | 17

3. Secondary Outcome: Infants: Percentages of Participants With RSV LRTI With Hospitalization From Delivery
Description: Percentages of infants with RSV LRTI with hospitalization from delivery through 90, 120, 150, and 180 days of life.
Time Frame: Delivery to 180 days after delivery
Population: The analysis population includes infant participants who were ≥ 37 weeks GA at birth and born to maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery, and had not received prophylactic treatment with palivizumab between birth and Day 180 after delivery, and had at least 1 documented post-partum contact during which active and/or passive surveillance activities for RSV-suspect illness could occur.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 2765 | 1430
Participants
  Day 90 | 57 | 53
  Day 120 | 64 | 56
  Day 150 | 67 | 57
  Day 180 | 68 | 59

4. Secondary Outcome: Infant: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Neonatal Period and Through the First Year of Life
Description: Number of infants with AEs and SAEs (with special attention to congenital anomalies; respiratory failure other than RSV-associated hospitalization; neonatal death; infant death; sudden infant death syndrome; asphyxia; neonatal or hypoxic-ischemic encephalopathy; or other adverse events or complications of adverse events that necessitate hospitalization) during the neonatal period and through the first year of life.
Time Frame: Delivery to 364 days after delivery
Population: The analysis population includes all infants born live to maternal subjects who received any test article and was analyzed as randomized unless conclusive documentation existed to confirm the mis-dosing of their respective mother and the identity of the treatment actually received.
Measure: Number; unit: participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
participants
  Any AEs | 2468 | 1295
  Overall SAEs (Including AESIs) | 1337 | 724
  Pre-Specified AESIs | 275 | 151

5. Secondary Outcome: Infants: Number of Participants With Potential Developmental Delay
Description: Number of infants with potential developmental delay (a term used to describe a delay in a child's development), as measured by the outcome of testing with the Ages and Stages Questionnaire-3 at 6 months and at 1 year, in infants of RSV F vaccinees as compared to placebo.
Time Frame: Day 180 after delivery
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
participants
  With any 6 months ASQ data | 2835 | 1460
  On schedule for communication | 2773 | 1424
  On schedule for Gross Motor | 2588 | 1298
  On schedule for Fine Motor | 2603 | 1364
  On schedule for Problem Solving | 2648 | 1381
  On Schedule for Personal-Social | 2481 | 1280

6. Secondary Outcome: Maternal: Number of Participants With Solicited Injection Site and Systemic Reactogenicity
Description: A number of maternal participants with solicited injection site and systemic reactogenicity within seven days of vaccination.
Time Frame: Day 0 to Day 7
Population: The analysis population includes maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery.
Measure: Number; unit: participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3045 | 1581
participants
  Total Solicited Local AE's | 1240 | 157
  Total Solicited Systematic AE's | 1255 | 611

7. Secondary Outcome: Maternal: Number of Participants With Unsolicited Adverse Events, Medically-attended Adverse Events (MAEs), Significant New Medical Conditions (SNMCs) and Serious Adverse Events (SAEs)
Description: Number of maternal participants with unsolicited (local and systemic) adverse events (AEs), unscheduled medically-attended adverse events (MAEs), significant new medical conditions (SNMCs), and serious adverse events (SAEs) through delivery and six (6) months thereafter.
Time Frame: Delivery to 180 days after delivery
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3045 | 1581
participants
  Unsolicited AEs | 2004 | 1022
  MAEs | 1534 | 802
  SNMCs | 65 | 38
  SAEs | 906 | 455

8. Secondary Outcome: Maternal: Number of Participants With Caesarean, Vaginal, or Instrument Assisted Vaginal Modes of Delivery
Description: Number of maternal subjects that had either Caesarean, vaginal, or instrument-assisted vaginal modes of delivery.
Time Frame: Delivery
Population: as for outcome 6
Measure: Number; unit: count of participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3045 | 1581
count of participants
  No Data | 22 | 16
  Vaginal (spontaneous) | 2110 | 1076
  Forceps or vacuum assisted delivery | 91 | 56
  Planned (repeat) Caesarean delivery | 225 | 132
  Planned (primary) Caesarean delivery | 111 | 47
  Caesarean delivery after failed attempt at vaginal delivery | 123 | 66
  Emergency Caesarean delivery | 347 | 178
  Unknown | 16 | 10

9. Secondary Outcome: Maternal: Immunogenicity of RSV F Vaccine and Placebo Expressed as GMFR
Description: Immunogenicity of RSV F Vaccine and Placebo (Anti-F IgG, PCA, and RSV Types A and B - MN assays) among Maternal Participants from Day 14 until Delivery
Time Frame: Day 14 to Delivery
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Ratio
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 2775 | 1445
Fold Ratio
  Day 14 (Anti F-IgG): number analyzed (Participants) | 2641 | 1369
  Day 14 (Anti F-IgG) | 18.59 [17.85 to 19.37] | 0.99 [0.97 to 1.02]
  Delivery (Anti F-IgG) | 14.37 [13.86 to 14.90] | 0.92 [0.90 to 0.95]
  Day 14 (PCA): number analyzed (Participants) | 2642 | 1369
  Day 14 (PCA) | 12.38 [11.97 to 12.81] | 0.94 [0.92 to 0.96]
  Delivery (PCA) | 9.94 [9.64 to 10.25] | 0.92 [0.90 to 0.94]
  Day 14 (MN - RSV/A): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/A) | 2.35 [2.06 to 2.68] | 0.98 [0.92 to 1.05]
  Delivery (MN - RSV/A): number analyzed (Participants) | 877 | 489
  Delivery (MN - RSV/A) | 2.20 [2.10 to 2.30] | 0.89 [0.86 to 0.93]
  Day 14 (MN - RSV/B): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/B) | 3.00 [2.56 to 3.51] | 0.96 [0.88 to 1.04]
  Delivery (MN - RSV/B): number analyzed (Participants) | 876 | 489
  Delivery (MN - RSV/B) | 2.15 [2.06 to 2.25] | 0.88 [0.84 to 0.93]

10. Secondary Outcome: Maternal: Percentage of Participants With a Seroresponse to RSV F Vaccine and Placebo
Description: as for outcome 9
Time Frame: Day 14 to Delivery
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum): Maternal subjects were administered with the adjuvanted RSV F vaccine (120 µg RSV F protein adsorbed to a 0.4 mg dose of aluminum as the phosphate salt) as a single 0.5 mL IM injection into the deltoid muscle.
- Formulated Buffer (Placebo Control): Maternal subjects were administered with the formulated buffer (placebo control) as a single 0.5 mL IM injection into the deltoid muscle.
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3045 | 1581
percentage of participants
  Day 14 (Anti F-IgG): number analyzed (Participants) | 2641 | 1369
  Day 14 (Anti F-IgG) | 98.3 [97.7 to 98.7] | 5.0 [3.9 to 6.3]
  Delivery (Anti F-IgG): number analyzed (Participants) | 2775 | 1445
  Delivery (Anti F-IgG) | 97.5 [96.8 to 98.0] | 5.0 [3.9 to 6.2]
  Day 14 (PCA): number analyzed (Participants) | 2642 | 1369
  Day 14 (PCA) | 99.4 [99.0 to 99.7] | 5.0 [3.9 to 6.3]
  Delivery (PCA): number analyzed (Participants) | 2775 | 1445
  Delivery (PCA) | 97.9 [97.3 to 98.4] | 4.2 [3.2 to 5.4]
  Day 14 (MN - RSV/A): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/A) | 71.3 [61.0 to 80.1] | 4.3 [1.2 to 10.8]
  Delivery (MN - RSV/A): number analyzed (Participants) | 877 | 489
  Delivery (MN - RSV/A) | 55.6 [52.3 to 59.0] | 4.9 [3.2 to 7.2]
  Day 14 (MN - RSV/B): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/B) | 70.2 [59.9 to 79.2] | 8.7 [3.8 to 16.4]
  Delivery (MN - RSV/B): number analyzed (Participants) | 876 | 489
  Delivery (MN - RSV/B) | 57.2 [53.8 to 60.5] | 4.9 [3.2 to 7.2]

11. Secondary Outcome: Maternal: Percentage of Participants Who Seroconverted (2 Fold Increase) as Determined by Immunogenicity of RSV F Vaccine and Placebo
Description: as for outcome 9
Time Frame: Day 14 to Delivery
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3045 | 1581
percentage of participants
  Day 14 (Anti F-IgG): number analyzed (Participants) | 2641 | 1369
  Day 14 (Anti F-IgG) | 98.3 [97.8 to 98.8] | 1.1 [0.6 to 1.8]
  Delivery(Anti F-IgG): number analyzed (Participants) | 2775 | 1445
  Delivery(Anti F-IgG) | 98.1 [97.5 to 98.5] | 2.2 [1.5 to 3.1]
  Day 14 (PCA): number analyzed (Participants) | 2642 | 1369
  Day 14 (PCA) | 98.0 [97.3 to 98.5] | 0.5 [0.2 to 1.1]
  Delivery (PCA): number analyzed (Participants) | 2775 | 1445
  Delivery (PCA) | 97.7 [97.1 to 98.3] | 2.1 [1.4 to 3.0]
  Day 14 (MN - RSV/A): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/A) | 69.1 [58.8 to 78.3] | 4.3 [1.2 to 10.8]
  Delivery (MN - RSV/A): number analyzed (Participants) | 877 | 489
  Delivery (MN - RSV/A) | 59.0 [55.6 to 62.2] | 5.5 [3.7 to 7.9]
  Day 14 (MN - RSV/B): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/B) | 70.2 [59.9 to 79.2] | 8.7 [3.8 to 16.4]
  Delivery (MN - RSV/B): number analyzed (Participants) | 876 | 489
  Delivery (MN - RSV/B) | 53.2 [49.8 to 56.5] | 4.3 [2.7 to 6.5]

12. Secondary Outcome: Maternal: Percentage of Participants Who Seroconverted (4 Fold Increase) as Determined by Immunogenicity of RSV F Vaccine and Placebo
Description: as for outcome 9
Time Frame: Day 14 to Delivery
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3045 | 1581
percentage of participants
  Day 14 (Anti F-IgG): number analyzed (Participants) | 2641 | 1369
  Day 14 (Anti F-IgG) | 91.8 [90.7 to 92.8] | 0.4 [0.2 to 1.0]
  Delivery(Anti F-IgG): number analyzed (Participants) | 2775 | 1445
  Delivery(Anti F-IgG) | 89.7 [88.5 to 90.8] | 0.9 [0.5 to 1.5]
  Day 14 (PCA): number analyzed (Participants) | 2642 | 1369
  Day 14 (PCA) | 88.1 [86.8 to 89.3] | 0.2 [0.0 to 0.6]
  Delivery (PCA): number analyzed (Participants) | 2775 | 1445
  Delivery (PCA) | 84.8 [83.4 to 86.1] | 0.6 [0.3 to 1.2]
  Day 14 (MN - RSV/A): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/A) | 19.1 [11.8 to 28.6] | 0 [0.0 to 3.9]
  Delivery (MN - RSV/A): number analyzed (Participants) | 877 | 489
  Delivery (MN - RSV/A) | 18.6 [16.1 to 21.3] | 1.2 [0.5 to 2.7]
  Day 14 (MN - RSV/B): number analyzed (Participants) | 94 | 92
  Day 14 (MN - RSV/B) | 35.1 [25.5 to 45.6] | 1.1 [0.0 to 5.9]
  Delivery (MN - RSV/B): number analyzed (Participants) | 876 | 489
  Delivery (MN - RSV/B) | 17.6 [15.1 to 20.3] | 1.0 [0.3 to 2.4]

13. Secondary Outcome: Immunogenicity of RSV F Vaccine and Placebo Expressed as GMT
Description: Immunogenicity of RSV F Vaccine and Placebo (Anti-F IgG, PCA, and RSV Types A and B - MN assays) among Infant Participants from Delivery until Day 180
Time Frame: Delivery to Day 180
Population: The analysis population includes infant participants who were ≥ 37 weeks GA at birth and born to maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
percentage of participants
  Delivery (Anti-F IgG): number analyzed (Participants) | 2557 | 1342
  Delivery (Anti-F IgG) | 9501 [9224 to 9787] | 752 [719 to 786]
  Day 14 (Anti-F IgG): number analyzed (Participants) | 799 | 403
  Day 14 (Anti-F IgG) | 6465 [6134 to 6815] | 543 [502 to 588]
  Day 35 (Anti-F IgG): number analyzed (Participants) | 770 | 416
  Day 35 (Anti-F IgG) | 3883 [3683 to 4094] | 324 [304 to 346]
  Day 60 (Anti-F IgG): number analyzed (Participants) | 711 | 360
  Day 60 (Anti-F IgG) | 2355 [2230 to 2487] | 242 [231 to 254]
  Day 90 (Anti-F IgG): number analyzed (Participants) | 677 | 348
  Day 90 (Anti-F IgG) | 1298 [1220 to 1382] | 216 [209 to 224]
  Day 112/120 (Anti-F IgG): number analyzed (Participants) | 641 | 329
  Day 112/120 (Anti-F IgG) | 690 [645 to 737] | 218 [209 to 227]
  Day 180 (Anti-F IgG): number analyzed (Participants) | 619 | 293
  Day 180 (Anti-F IgG) | 289 [273 to 305] | 218 [209 to 227]
  Delivery (PCA): number analyzed (Participants) | 2547 | 1336
  Delivery (PCA) | 136 [132 to 139] | 15 [14 to 15]
  Day 14 (PCA): number analyzed (Participants) | 776 | 395
  Day 14 (PCA) | 103 [98 to 107] | 12 [11 to 12]
  Day 35 (PCA): number analyzed (Participants) | 759 | 406
  Day 35 (PCA) | 69 [66 to 72] | 8 [8 to 8]
  Day 60 (PCA): number analyzed (Participants) | 699 | 355
  Day 60 (PCA) | 45 [43 to 48] | 7 [6 to 7]
  Day 90 (PCA): number analyzed (Participants) | 666 | 343
  Day 90 (PCA) | 29 [27 to 30] | 6 [6 to 7]
  Day 112/120 (PCA): number analyzed (Participants) | 627 | 327
  Day 112/120 (PCA) | 17 [16 to 18] | 6 [6 to 7]
  Day 180 (PCA): number analyzed (Participants) | 615 | 291
  Day 180 (PCA) | 8 [8 to 9] | 6 [6 to 7]
  Delivery (MN - RSV/A): number analyzed (Participants) | 758 | 424
  Delivery (MN - RSV/A) | 1705 [1602 to 1813] | 732 [674 to 796]
  Day 14 (MN - RSV/A): number analyzed (Participants) | 197 | 97
  Day 14 (MN - RSV/A) | 1108 [983 to 1250] | 505 [427 to 596]
  Day 35 (MN - RSV/A): number analyzed (Participants) | 206 | 130
  Day 35 (MN - RSV/A) | 609 [546 to 679] | 266 [233 to 304]
  Day 60 (MN - RSV/A): number analyzed (Participants) | 215 | 111
  Day 60 (MN - RSV/A) | 370 [330 to 415] | 190 [164 to 222]
  Day 90 (MN - RSV/A): number analyzed (Participants) | 199 | 104
  Day 90 (MN - RSV/A) | 201 [178 to 228] | 109 [92 to 130]
  Day 112/120 (MN - RSV/A): number analyzed (Participants) | 187 | 119
  Day 112/120 (MN - RSV/A) | 110 [96 to 127] | 61 [51 to 73]
  Day 180 (MN - RSV/A): number analyzed (Participants) | 189 | 93
  Day 180 (MN - RSV/A) | 41 [35 to 49] | 26 [20 to 35]
  Delivery (MN - RSV/B): number analyzed (Participants) | 757 | 423
  Delivery (MN - RSV/B) | 1292 [1198 to 1393] | 607 [544 to 678]
  Day 14 (MN - RSV/B): number analyzed (Participants) | 24 | 21
  Day 14 (MN - RSV/B) | 1079 [642 to 1813] | 324 [201 to 521]
  Day 35 (MN - RSV/B): number analyzed (Participants) | 20 | 24
  Day 35 (MN - RSV/B) | 422 [243 to 732] | 195 [134 to 248]
  Day 60 (MN - RSV/B): number analyzed (Participants) | 18 | 19
  Day 60 (MN - RSV/B) | 216 [151 to 309] | 151 [82 to 279]
  Day 90 (MN - RSV/B): number analyzed (Participants) | 21 | 16
  Day 90 (MN - RSV/B) | 185 [113 to 301] | 61 [34 to 111]
  Day 112/120 (MN - RSV/B): number analyzed (Participants) | 13 | 25
  Day 112/120 (MN - RSV/B) | 71 [39 to 131] | 48 [31 to 73]
  Day 180 (MN - RSV/B): number analyzed (Participants) | 18 | 15
  Day 180 (MN - RSV/B) | 34 [17 to 65] | 24 [9 to 67]

14. Secondary Outcome: Infants: Percentage of Participants With a Seroresponse to RSV F Vaccine and Placebo
Description: as for outcome 13
Time Frame: Delivery to Day 180
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
percentage of participants
  Delivery (Anti-F IgG): number analyzed (Participants) | 2558 | 1342
  Delivery (Anti-F IgG) | 95.9 [95.1 to 96.7] | 5.0 [3.9 to 6.3]
  Day 14 (Anti-F IgG): number analyzed (Participants) | 810 | 409
  Day 14 (Anti-F IgG) | 95.9 [94.3 to 97.2] | 4.9 [3.0 to 7.5]
  Day 35 (Anti-F IgG): number analyzed (Participants) | 802 | 439
  Day 35 (Anti-F IgG) | 94.1 [92.3 to 95.7] | 4.8 [3.0 to 7.2]
  Day 60 (Anti-F IgG): number analyzed (Participants) | 778 | 410
  Day 60 (Anti-F IgG) | 94.2 [92.3 to 95.8] | 4.9 [3.0 to 7.4]
  Day 90 (Anti-F IgG): number analyzed (Participants) | 805 | 411
  Day 90 (Anti-F IgG) | 77.0 [74.0 to 79.9] | 4.9 [3.0 to 7.4]
  Day 112/120 (Anti-F IgG): number analyzed (Participants) | 766 | 409
  Day 112/120 (Anti-F IgG) | 36.4 [33.0 to 39.9] | 4.9 [3.0 to 7.5]
  Day 180 (Anti-F IgG): number analyzed (Participants) | 770 | 388
  Day 180 (Anti-F IgG) | 6.5 [4.9 to 8.5] | 4.9 [3.0 to 7.5]
  Delivery (PCA): number analyzed (Participants) | 2548 | 1336
  Delivery (PCA) | 96.8 [96.0 to 97.4] | 4.6 [3.5 to 5.8]
  Day 14 (PCA): number analyzed (Participants) | 787 | 401
  Day 14 (PCA) | 95.4 [93.7 to 96.8] | 4.7 [2.9 to 7.3]
  Day 35 (PCA): number analyzed (Participants) | 791 | 429
  Day 35 (PCA) | 95.6 [93.9 to 96.9] | 4.4 [2.7 to 6.8]
  Day 60 (PCA): number analyzed (Participants) | 766 | 405
  Day 60 (PCA) | 92.0 [89.9 to 93.9] | 4.4 [2.7 to 6.9]
  Day 90 (PCA): number analyzed (Participants) | 793 | 406
  Day 90 (PCA) | 73.1 [69.9 to 76.2] | 4.7 [2.8 to 7.2]
  Day 112/120 (PCA): number analyzed (Participants) | 751 | 406
  Day 112/120 (PCA) | 29.7 [26.4 to 33.1] | 4.7 [2.8 to 7.2]
  Day 180 (PCA): number analyzed (Participants) | 762 | 386
  Day 180 (PCA) | 5.2 [3.8 to 7.1] | 4.1 [2.4 to 6.6]
  Delivery (MN - RSV/A): number analyzed (Participants) | 758 | 424
  Delivery (MN - RSV/A) | 20.2 [17.4 to 23.2] | 5.0 [3.1 to 7.5]
  Day 14 (MN - RSV/A): number analyzed (Participants) | 197 | 98
  Day 14 (MN - RSV/A) | 14.2 [9.7 to 19.9] | 3.1 [0.6 to 8.7]
  Day 35 (MN - RSV/A): number analyzed (Participants) | 215 | 137
  Day 35 (MN - RSV/A) | 19.5 [14.5 to 25.5] | 3.6 [1.2 to 8.3]
  Day 60 (MN - RSV/A): number analyzed (Participants) | 230 | 125
  Day 60 (MN - RSV/A) | 17.4 [12.7 to 22.9] | 4.8 [1.8 to 10.2]
  Day 90 (MN - RSV/A): number analyzed (Participants) | 225 | 125
  Day 90 (MN - RSV/A) | 13.8 [9.6 to 19.0] | 4.8 [1.8 to 10.2]
  Day 112/120 (MN - RSV/A): number analyzed (Participants) | 221 | 141
  Day 112/120 (MN - RSV/A) | 8.6 [5.3 to 13.1] | 5.0 [2.0 to 10.0]
  Day 180 (MN - RSV/A): number analyzed (Participants) | 229 | 118
  Day 180 (MN - RSV/A) | 3.5 [1.5 to 6.8] | 4.2 [1.4 to 9.6]
  Delivery (MN - RSV/B): number analyzed (Participants) | 757 | 423
  Delivery (MN - RSV/B) | 11.2 [9.1 to 13.7] | 4.3 [2.5 to 6.6]
  Day 14 (MN - RSV/B): number analyzed (Participants) | 24 | 22
  Day 14 (MN - RSV/B) | 54.2 [32.8 to 74.4] | 4.5 [0.1 to 22.8]
  Day 35 (MN - RSV/B): number analyzed (Participants) | 22 | 24
  Day 35 (MN - RSV/B) | 27.3 [10.7 to 50.2] | 4.2 [0.1 to 21.1]
  Day 60 (MN - RSV/B): number analyzed (Participants) | 20 | 24
  Day 60 (MN - RSV/B) | 5.0 [0.1 to 24.9] | 4.2 [0.1 to 21.1]
  Day 90 (MN - RSV/B): number analyzed (Participants) | 25 | 24
  Day 90 (MN - RSV/B) | 40.0 [21.1 to 61.3] | 4.2 [0.1 to 21.1]
  Day 112/120 (MN - RSV/B): number analyzed (Participants) | 19 | 27
  Day 112/120 (MN - RSV/B) | 5.3 [0.1 to 26.0] | 3.7 [0.1 to 19.0]
  Day 180 (MN - RSV/B): number analyzed (Participants) | 22 | 23
  Day 180 (MN - RSV/B) | 4.5 [0.1 to 22.8] | 4.3 [0.1 to 21.9]

15. Secondary Outcome: Infant: Immunogenicity of RSV F Vaccine and Placebo Expressed as GMR
Description: Immunogenicity of RSV F Vaccine and Placebo (Anti-F IgG, PCA, and RSV Types A and B - MN assays) among Infant Participants from Day 14 until Day 180
Time Frame: Day 14 to Day 180
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Ratio
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
Fold Ratio
  Day 14 (Anti-F IgG): number analyzed (Participants) | 810 | 408
  Day 14 (Anti-F IgG) | 0.67 [0.65 to 0.69] | 0.69 [0.65 to 0.72]
  Day 35 (Anti-F IgG): number analyzed (Participants) | 802 | 439
  Day 35 (Anti-F IgG) | 0.42 [0.41 to 0.43] | 0.44 [0.42 to 0.47]
  Day 60 (Anti-F IgG): number analyzed (Participants) | 777 | 410
  Day 60 (Anti-F IgG) | 0.24 [0.24 to 0.25] | 0.35 [0.33 to 0.35]
  Day 90 (Anti-F IgG): number analyzed (Participants) | 805 | 410
  Day 90 (Anti-F IgG) | 0.13 [0.13 to 0.14] | 0.30 [0.28 to 0.33]
  Day 112/120 (Anti-F IgG): number analyzed (Participants) | 766 | 409
  Day 112/120 (Anti-F IgG) | 0.07 [0.07 to 0.08] | 0.33 [0.29 to 0.36]
  Day 180 (Anti-F IgG): number analyzed (Participants) | 769 | 388
  Day 180 (Anti-F IgG) | 0.03 [0.03 to 0.03] | 0.32 [0.29 to 0.36]
  Day 14 (PCA): number analyzed (Participants) | 784 | 400
  Day 14 (PCA) | 0.76 [0.73 to 0.78] | 0.76 [0.74 to 0.79]
  Day 35 (PCA): number analyzed (Participants) | 790 | 427
  Day 35 (PCA) | 0.51 [0.49 to 0.52] | 0.58 [0.55 to 0.60]
  Day 60 (PCA): number analyzed (Participants) | 766 | 405
  Day 60 (PCA) | 0.34 [0.33 to 0.35] | 0.49 [0.46 to 0.53]
  Day 90 (PCA): number analyzed (Participants) | 790 | 404
  Day 90 (PCA) | 0.21 [0.20 to 0.22] | 0.46 [0.42 to 0.49]
  Day 112/120 (PCA): number analyzed (Participants) | 749 | 403
  Day 112/120 (PCA) | 0.12 [0.12 to 0.13] | 0.51 [0.47 to 0.56]
  Day 180 (PCA): number analyzed (Participants) | 761 | 385
  Day 180 (PCA) | 0.06 [0.06 to 0.06] | 0.50 [0.46 to 0.54]
  Day 14 (MN - RSV/A): number analyzed (Participants) | 192 | 95
  Day 14 (MN - RSV/A) | 0.68 [0.64 to 0.72] | 0.69 [0.63 to 0.75]
  Day 35 (MN - RSV/A): number analyzed (Participants) | 203 | 128
  Day 35 (MN - RSV/A) | 0.39 [0.36 to 0.42] | 0.40 [0.37 to 0.43]
  Day 60 (MN - RSV/A): number analyzed (Participants) | 216 | 117
  Day 60 (MN - RSV/A) | 0.21 [0.20 to 0.23] | 0.27 [0.25 to 0.30]
  Day 90 (MN - RSV/A): number analyzed (Participants) | 214 | 121
  Day 90 (MN - RSV/A) | 0.13 [0.12 to 0.14] | 0.17 [0.15 to 0.19]
  Day 112/120 (MN - RSV/A): number analyzed (Participants) | 207 | 132
  Day 112/120 (MN - RSV/A) | 0.08 [0.07 to 0.09] | 0.10 [0.09 to 0.12]
  Day 180 (MN - RSV/A): number analyzed (Participants) | 215 | 112
  Day 180 (MN - RSV/A) | 0.03 [0.02 to 0.03] | 0.05 [0.04 to 0.07]
  Day 14 (MN - RSV/B): number analyzed (Participants) | 24 | 21
  Day 14 (MN - RSV/B) | 0.55 [0.48 to 0.65] | 0.66 [0.57 to 0.76]
  Day 35 (MN - RSV/B): number analyzed (Participants) | 22 | 24
  Day 35 (MN - RSV/B) | 0.39 [0.31 to 0.50] | 0.34 [0.28 to 0.40]
  Day 60 (MN - RSV/B): number analyzed (Participants) | 20 | 24
  Day 60 (MN - RSV/B) | 0.17 [0.12 to 0.23] | 0.22 [0.16 to 0.29]
  Day 90 (MN - RSV/B): number analyzed (Participants) | 25 | 24
  Day 90 (MN - RSV/B) | 0.11 [0.07 to 0.15] | 0.16 [0.11 to 0.24]
  Day 112/120 (MN - RSV/B): number analyzed (Participants) | 19 | 27
  Day 112/120 (MN - RSV/B) | 0.07 [0.05 to 0.08] | 0.08 [0.06 to 0.12]
  Day 180 (MN - RSV/B): number analyzed (Participants) | 22 | 23
  Day 180 (MN - RSV/B) | 0.03 [0.01 to 0.05] | 0.05 [0.03 to 0.08]

16. Secondary Outcome: Infants: Mean Length of Participants at Birth
Description: Length of Infant participants measured at delivery expressed in centimeters
Time Frame: At Delivery
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
centimeters | 50.04 (2.921) | 50.16 (3.144)

17. Secondary Outcome: Infants: Mean Weight of Participants at Birth
Description: Weight of infant participants measured at delivery expressed in kilograms.
Time Frame: At Delivery
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
kg | 3.21 (0.484) | 3.20 (0.505)

18. Secondary Outcome: Infants: Mean Frontal-occipital Head Circumference of Participants at Birth
Description: Frontal-occipital Head Circumference measured in infant participants at delivery expressed as centimeters
Time Frame: At Delivery
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
centimeters | 34.2 (2.08) | 34.2 (1.77)

19. Secondary Outcome: Infants: Mean APGAR (Appearance, Pulse, Grimace, Activity, Respiration) Score of Participants at Birth
Description: The APGAR test measures the infant's Appearance, Pulse, Grimace, Activity, and Respiration. Any score of 7 or above is considered a good APGAR score.
  The maximum APGAR score is 10 and the minimum score is 1.
Time Frame: At Delivery
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
units on a scale
  1 minute | 8.4 (1.08) | 8.4 (1.17)
  5 minute | 9.4 (0.78) | 9.4 (0.91)

20. Secondary Outcome: Maternal: Number of Participants With Post-immunization Onset of Specific Complications of Third-trimester Pregnancy and Delivery
Description: Number of maternal participants with post-immunization onset of specific complications of third-trimester pregnancy and delivery including Pregnancy complications, Labor and delivery complications.
Time Frame: Day 0 to Delivery
Population: maternal safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3045 | 1581
Participants
  No | 2528 | 1295
  Yes | 488 | 268
  No Data | 13 | 8
  Subjects without delivery data | 16 | 10

21. Secondary Outcome: Infants: Number of Participants With Developmental Delay
Description: Number of infants with developmental delay (a term used to describe a delay in a child's development.), as measured by the outcome of testing at 1 year, in infants of RSV F vaccinees as compared to placebo.
Time Frame: Day 364 after delivery
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 3008 | 1561
participants
  With any 12 months ASQ data | 2707 | 1395
  On schedule for communication | 2670 | 1387
  On schedule for Gross Motor | 2535 | 1318
  On schedule for Fine Motor | 2535 | 1318
  On schedule for Problem Solving | 2546 | 1325
  On Schedule for Personal-Social | 2559 | 1317

22. Secondary Outcome: Maternal: Immunogenicity of Anti-RSV F IgG and Placebo Expressed as GMEU (Geometric Mean ELISA Units/mL)
Description: Immunogenicity of RSV F Vaccine and Placebo (Anti-F IgG) among Maternal Participants from Screening until Delivery
Time Frame: Pre-dose to Delivery +180 days
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EU (ELISA units/mL)
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 2775 | 1445
EU (ELISA units/mL)
  Pre-Dose | 568 [551 to 586] | 569 [546 to 594]
  Day 14: number analyzed (Participants) | 2641 | 1369
  Day 14 | 10568 [10249 to 10897] | 563 [539 to 587]
  Delivery | 8164 [7944 to 8390] | 525 [504 to 547]

23. Secondary Outcome: Maternal: Immunogenicity of RSV F Vaccine and Placebo Expressed as GMC (Geometric Mean Concentration)
Description: Immunogenicity of RSV F Vaccine and Placebo (Palivizumab-competitive antibodies (PCA)) among Maternal Participants from Screening until Delivery
Time Frame: Pre-dose to Delivery +180 days
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 2775 | 1445
µg/mL
  Pre-Dose | 13 [13 to 13] | 13 [13 to 14]
  Day 14: number analyzed (Participants) | 2642 | 1369
  Day 14 | 162 [158 to 167] | 13 [12 to 13]
  Delivery | 130 [127 to 133] | 12 [12 to 13]

24. Secondary Outcome: Maternal: Immunogenicity of RSV F Vaccine and Placebo Expressed as GMT (Geometric Mean Titers)
Description: Immunogenicity of RSV F Vaccine and Placebo (RSV/A microneutralization titers expressed as GMT) among Maternal Participants from Screening until Delivery
Time Frame: Pre-dose to Delivery +180 days
Population: The analysis population includes maternal participants who received a study injection as randomized and ≥ 2 weeks prior to delivery.
  Per-Protocol Immunogenicity Maternal (PP-IMM-M) participant population is analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 879 | 489
titers
  Pre-Dose | 714 [677 to 753] | 741 [691 to 794]
  Day 14 | 1622 [1384 to 1900] | 654 [565 to 756]
  Delivery | 1569 [1488 to 1654] | 663 [616 to 713]

25. Secondary Outcome: Maternal: Immunogenicity of RSV F Vaccine and Placebo Expressed as GMTs
Description: Immunogenicity of RSV F Vaccine and Placebo (RSV/B microneutralization titers expressed as GMT) among Maternal Participants from Screening until Delivery
Time Frame: Pre-dose to Delivery +180 days
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Formulated Buffer (Placebo Control)
Number analyzed (Participants) | 879 | 489
titers
  Pre-Dose | 563 [525 to 605] | 605 [552 to 664]
  Day 14 | 2419 [1934 to 3025] | 845 [670 to 1066]
  Delivery | 1213 [1138 to 1293] | 534 [487 to 586]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious Adverse Events Other (Not Including Serious) Adverse Events
Groups:
- Maternal ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum): Maternal participants were administered with the adjuvanted RSV F vaccine 120 µg RSV F protein adsorbed to a 0.4 mg dose of aluminum (as the phosphate salt) as a single 0.5 mL IM injection into the deltoid muscle.
- Maternal ; Formulated Buffer (Placebo Control): Maternal participants were administered with the formulated buffer (placebo control) as a single 0.5 mL IM injection into the deltoid muscle.
- Infant ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum): Infants in which mother received RSV F vaccine 120 µg RSV F protein adsorbed to a 0.4 mg dose of aluminum (as the phosphate salt) as a single 0.5 mL IM injection into the deltoid muscle..
- Infant ; Formulated Buffer (Placebo Control): Infants in which mother received formulated buffer (placebo control) as a single 0.5 mL IM injection into the deltoid muscle.
Arm/Group | Maternal ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Maternal ; Formulated Buffer (Placebo Control) | Infant ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) | Infant ; Formulated Buffer (Placebo Control)
All-Cause Mortality (participants affected / at risk) | 0/3045 | 0/1581 | 0/3008 | 0/1561
Serious Adverse Events (participants affected / at risk) | 1356/3045 | 684/1581 | 2535/3008 | 1396/1561
Other Adverse Events (participants affected / at risk) | 361/4636 | 185/4636 | 3167/4569 | 1598/4569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Maternal ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) (N=3045) | Maternal ; Formulated Buffer (Placebo Control) (N=1581) | Infant ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) (N=3008) | Infant ; Formulated Buffer (Placebo Control) (N=1561)
Anaemia (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Anaemia neonatal (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Polycythaemia neonatorum (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Bradycardia neonatal (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Cyanosis (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Neonatal tachycardia (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Right atrial dilatation (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
ABO haemolytic disease of newborn (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Abnormal palmar/plantar creases (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 6 (6) | 3 (3)
Accessory auricle (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 10 (10) | 1 (1)
Accessory breast (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Anal atresia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 44 (45) | 19 (19)
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Anomaly of external ear congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 7 (9) | 7 (8)
Beckwith-Wiedemann syndrome (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Birth mark (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 195 (199) | 96 (99)
Branchial cyst (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Buried penis syndrome (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Camptodactyly congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Cardiac septal defect (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Cataract congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cerebral palsy (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Choledochal cyst (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Chondrodystrophy (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Chordee (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Chromosomal deletion (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cleft lip (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Cleft palate (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Cleft uvula (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Clinodactyly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 6 (6) | 1 (1)
Congenital acrochordon (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 13 (13) | 4 (4)
Congenital aortic anomaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital cerebral cyst (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital claw toe (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital cleft hand (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital eye disorder (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital genital malformation female (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Congenital hearing disorder (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital hyperextension of knee (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 1 (1)
Congenital knee dislocation (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Congenital megacolon (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Congenital melanocytic naevus (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 12 (13) | 1 (1)
Congenital melanosis (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 9 (9) | 2 (2)
Congenital mitral valve incompetence (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital naevus (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 307 (314) | 177 (183)
Congenital nephrotic syndrome (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital nose malformation (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Congenital pneumonia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 7 (7) | 3 (3)
Congenital pulmonary artery anomaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital pulmonary hypertension (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Congenital renal disorder (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 22 (22) | 14 (14)
Congenital torticollis (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 5 (5)
Congenital tracheomalacia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital tricuspid valve incompetence (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 261 (261) | 146 (146)
Congenital varicella infection (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Congenital vesicoureteric reflux (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 4 (4)
Cryptorchism (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 10 (11) | 7 (7)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 3 (3)
Deafness congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 3 (4) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 4 (4)
Ear malformation (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Extrarenal pelvis (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Eyelid ptosis congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Galactosaemia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 2 (2)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 24 (27) | 23 (25)
Heart disease congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Heterochromia iridis (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 19 (19) | 4 (4)
Hypertelorism of orbit (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 1 (1)
Interruption of aortic arch (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Intestinal malrotation (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Labial tie (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 5 (5)
Laryngomalacia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 6 (7) | 5 (5)
Low set ears (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Macrocephaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 4 (5)
Macroglossia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Microcephaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 23 (24) | 9 (9)
Micrognathia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Microtia (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Mosaicism (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Naevus flammeus (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 17 (17) | 5 (5)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 2 (2)
Pectus excavatum (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Penile torsion (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 0 (0)
Persistent foetal circulation (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 4 (4)
Persistent pupillary membrane (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Pilonidal cyst congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Plagiocephaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 4 (4)
Polydactyly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 16 (16) | 7 (7)
Preauricular cyst (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 6 (6)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Scaphocephaly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Sebaceous naevus (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 2 (2)
Single umbilical artery (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Skull malformation (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Strabismus congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 7 (7) | 1 (1)
Supernumerary nipple (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 6 (6) | 4 (4)
Syndactyly (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 1 (1)
Telangiectasia congenital (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Thalassaemia alpha (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (2)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 5 (6)
Conductive deafness (Ear and labyrinth disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Opsoclonus myoclonus (Eye disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 17 (18) | 4 (4)
Enterocolitis (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Infantile vomiting (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Neonatal intestinal dilatation (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 2 (2)
Death (General disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 1 (1)
Death neonatal (General disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 3 (3)
Developmental delay (General disorders) | 0/0 (0) | 0/0 (0) | 10 (10) | 2 (2)
Fever neonatal (General disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 1 (1)
Macrosomia (General disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 2 (2)
Sudden infant death syndrome (General disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Temperature regulation disorder (General disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0/0 (0) | 0/0 (0) | 26 (26) | 11 (11)
Food allergy (Immune system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Adenovirus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 2 (2)
Bacterial sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (2)
Beta haemolytic streptococcal infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Bronchiolitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 85 (95) | 49 (52)
Bronchitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 6 (6) | 2 (3)
Cellulitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Corona virus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Eczema infected (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 50 (52) | 32 (34)
Gastroenteritis adenovirus (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Group B streptococcus neonatal sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0/0 (0) | 0/0 (0) | 3 (3) | 3 (3)
Klebsiella sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Listeria sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 17 (18) | 8 (8)
Lower respiratory tract infection viral (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Meningitis enteroviral (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 3 (3)
Meningitis neonatal (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Neonatal infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Neonatal pneumonia (Infections and infestations) | 0/0 (0) | 0/0 (0) | 11 (11) | 9 (9)
Nosocomial infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Omphalitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Ophthalmia neonatorum (Infections and infestations) | 0/0 (0) | 0/0 (0) | 4 (4) | 2 (2)
Oral candidiasis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Otitis media acute (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0/0 (0) | 0/0 (0) | 66 (72) | 70 (74)
Pneumonia viral (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 4 (4)
Pulmonary tuberculosis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 4 (4) | 6 (6)
Pyelonephritis acute (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 8 (8) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 8 (8) | 5 (5)
Respiratory tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 5 (5) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 4 (4) | 1 (1)
Rocky mountain spotted fever (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 2 (2)
Sepsis neonatal (Infections and infestations) | 0/0 (0) | 0/0 (0) | 43 (44) | 29 (29)
Septic rash (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Skin candida (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Tuberculosis of intrathoracic lymph nodes (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Umbilical sepsis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 12 (12) | 2 (2)
Urinary tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 15 (15) | 14 (14)
Urinary tract infection bacterial (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (3) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Varicella (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Injury to brachial plexus due to birth trauma (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Acoustic stimulation tests abnormal (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Apgar score low (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Body height below normal (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0/0 (0) | 0/0 (0) | 23 (23) | 13 (13)
Cardiac murmur functional (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
HIV test positive (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Haemoglobin abnormal (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Karyotype analysis abnormal (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Opiates positive (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Reflex test abnormal (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Vascular resistance pulmonary increased (Investigations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Cow's milk intolerance (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 14 (14) | 8 (8)
Failure to thrive (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 6 (6) | 3 (3)
Feeding intolerance (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 13 (13) | 13 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 2 (2)
Poor feeding infant (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 1 (1)
Underweight (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cranial sutures widening (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 4 (4)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Head deformity (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Joint laxity (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Positional plagiocephaly (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 0 (0)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Benign intracranial hypertension (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Convulsion neonatal (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Encephalopathy neonatal (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 7 (7) | 1 (1)
Epilepsy (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 0 (0)
Fine motor delay (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Gross motor delay (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 12 (12) | 7 (7)
Infantile spasms (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Poor sucking reflex (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Reflexes abnormal (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 2 (3) | 0 (0)
Status epilepticus (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Tethered cord syndrome (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 4 (4) | 2 (2)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 16 (16) | 8 (8)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 97 (98) | 52 (52)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 12 (12) | 3 (3)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 149 (149) | 98 (98)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Poor weight gain neonatal (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 151 (151) | 72 (72)
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 4 (4) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 2 (2)
Micturition frequency decreased (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (2) | 0 (0)
Renal failure neonatal (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Sterile pyuria (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Enlarged clitoris (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Neonatal testicular torsion (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Penis disorder (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Testicular retraction (Reproductive system and breast disorders) | 0/0 (0) | 0/0 (0) | 7 (8) | 5 (5)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (4)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 6 (8) | 3 (3)
Choking (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cyanosis neonatal (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Grunting (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 3 (3)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 16 (16) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 15 (15) | 10 (11)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 1 (1)
Neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 62 (62) | 36 (36)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 5 (5) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (3) | 2 (2)
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 19 (19) | 9 (9)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 28 (31) | 12 (12)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Eczema infantile (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Ephelides (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 17 (17) | 7 (7) | 0/0 (0) | 0/0 (0)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0/0 (0) | 0/0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0/0 (0) | 0/0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0/0 (0) | 0/0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Bradycardia foetal (Cardiac disorders) | 10 (10) | 3 (3) | 0/0 (0) | 0/0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0)
Foetal heart rate disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 24 (24) | 10 (10) | 0/0 (0) | 0/0 (0)
Tachycardia (Cardiac disorders) | 7 (7) | 4 (4) | 0/0 (0) | 0/0 (0)
Tachycardia foetal (Cardiac disorders) | 6 (6) | 5 (5) | 0/0 (0) | 0/0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0/0 (0) | 0/0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0/0 (0) | 0/0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 5 (5) | 1 (1) | 0/0 (0) | 0/0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Amniotic cavity infection (Infections and infestations) | 17 (17) | 12 (13) | 0/0 (0) | 0/0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0/0 (0) | 0/0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Breast abscess (Infections and infestations) | 5 (5) | 0 (0) | 0/0 (0) | 0/0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Cervicitis (Infections and infestations) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Endometritis (Infections and infestations) | 6 (6) | 3 (3) | 0/0 (0) | 0/0 (0)
Endometritis decidual (Infections and infestations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Funisitis (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 0/0 (0) | 0/0 (0)
HIV infection (Infections and infestations) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 0/0 (0) | 0/0 (0)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Mastitis (Infections and infestations) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Mastitis postpartum (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Postoperative wound infection (Infections and infestations) | 1 (2) | 3 (3) | 0/0 (0) | 0/0 (0)
Postpartum sepsis (Infections and infestations) | 8 (8) | 0 (0) | 0/0 (0) | 0/0 (0)
Puerperal pyrexia (Infections and infestations) | 4 (4) | 1 (1) | 0/0 (0) | 0/0 (0)
Pyelonephritis (Infections and infestations) | 5 (5) | 1 (1) | 0/0 (0) | 0/0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Sepsis (Infections and infestations) | 5 (5) | 1 (1) | 0/0 (0) | 0/0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Urinary tract infection (Infections and infestations) | 13 (13) | 10 (10) | 0/0 (0) | 0/0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Wound infection (Infections and infestations) | 1 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 5 (5) | 0/0 (0) | 0/0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Failed forceps delivery (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 0/0 (0) | 0/0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Uterine cervical laceration (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0/0 (0) | 0/0 (0)
Uterine dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Uterine rupture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0)
Vaginal laceration (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0/0 (0) | 0/0 (0)
Amniotic fluid index decreased (Investigations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Blood pressure increased (Investigations) | 3 (3) | 2 (2) | 0/0 (0) | 0/0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Foetal biophysical profile score abnormal (Investigations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Foetal heart rate increased (Investigations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Foetal monitoring abnormal (Investigations) | 5 (5) | 3 (3) | 0/0 (0) | 0/0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Seroconversion test positive (Investigations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Ultrasound Doppler abnormal (Investigations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Cervix warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 23 (23) | 6 (6) | 0/0 (0) | 0/0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 8 (8) | 0/0 (0) | 0/0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 47 (47) | 20 (20) | 0/0 (0) | 0/0 (0)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 6 (6) | 0/0 (0) | 0/0 (0)
Face presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 28 (28) | 11 (11) | 0/0 (0) | 0/0 (0)
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 0/0 (0) | 0/0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 200 (200) | 97 (97) | 0/0 (0) | 0/0 (0)
Foetal growth abnormality (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 4 (4) | 0/0 (0) | 0/0 (0)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 1 (1) | 0/0 (0) | 0/0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 4 (4) | 0/0 (0) | 0/0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 141 (142) | 66 (66) | 0/0 (0) | 0/0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0/0 (0) | 0/0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 7 (7) | 0/0 (0) | 0/0 (0)
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Induced labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Labour pain (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Maternal distress during labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0/0 (0) | 0/0 (0)
Meconium stain (Pregnancy, puerperium and perinatal conditions) | 16 (16) | 6 (6) | 0/0 (0) | 0/0 (0)
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 2 (2) | 0/0 (0) | 0/0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 4 (4) | 0/0 (0) | 0/0 (0)
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0) | 0/0 (0) | 0/0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Placental disorder (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Postmature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 35 (35) | 17 (17) | 0/0 (0) | 0/0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 72 (73) | 43 (43) | 0/0 (0) | 0/0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 174 (174) | 90 (90) | 0/0 (0) | 0/0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 12 (13) | 7 (9) | 0/0 (0) | 0/0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 24 (24) | 19 (19) | 0/0 (0) | 0/0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 7 (7) | 0/0 (0) | 0/0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 2 (2) | 0/0 (0) | 0/0 (0)
Previous caesarean section (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 81 (81) | 47 (47) | 0/0 (0) | 0/0 (0)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 23 (23) | 15 (15) | 0/0 (0) | 0/0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 14 (14) | 0/0 (0) | 0/0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 0/0 (0) | 0/0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0/0 (0) | 0/0 (0)
Retroplacental haematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 8 (8) | 0/0 (0) | 0/0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 0/0 (0) | 0/0 (0)
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Uterine hyperstimulation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 0/0 (0) | 0/0 (0)
Uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Conversion disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Perinatal depression (Psychiatric disorders) | 3 (3) | 2 (2) | 0/0 (0) | 0/0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0) | 0/0 (0) | 0/0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Shortened cervix (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Uterine atony (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Varicose veins vulval (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vulval haematoma (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Vulval oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0/0 (0) | 0/0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Hypertension (Vascular disorders) | 11 (11) | 6 (6) | 0/0 (0) | 0/0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Maternal ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) (N=4636) | Maternal ; Formulated Buffer (Placebo Control) (N=4636) | Infant ; Adjuvanted RSV F Vaccine (120 µg RSVF Protein Adsorbed to a 0.4 mg Dose of Aluminum) (N=4569) | Infant ; Formulated Buffer (Placebo Control) (N=4569)
Diarrhoea neonatal (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 252/3008 (312) | 115/1561 (137)
Vomiting (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 169/3008 (211) | 83/1561 (92)
Fever neonatal (General disorders) | 0/0 (0) | 0/0 (0) | 401/3008 (527) | 173/1561 (226)
Gastroenteritis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 182/3008 (211) | 84/1561 (88)
Ophthalmia neonatorum (Infections and infestations) | 0/0 (0) | 0/0 (0) | 195/3008 (213) | 97/1561 (109)
Oral candidiasis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 158/3008 (173) | 74/1561 (92)
Otitis media (Infections and infestations) | 0/0 (0) | 0/0 (0) | 159/3008 (205) | 94/1561 (126)
Upper respiratory tract infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 367/3008 (478) | 198/1561 (264)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 182/3008 (186) | 104/1561 (105)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 244/3008 (290) | 109/1561 (123)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 424/3008 (520) | 206/1561 (241)
Eczema infantile (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 231/3008 (245) | 126/1561 (137)
Rash (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0) | 203/3008 (246) | 135/1561 (152)
Headache (Nervous system disorders) | 361/3045 (458) | 185/1581 (221) | 0/0 (0) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT02624947/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT02624947/SAP_001.pdf